CLINICAL TRIAL: NCT03073655
Title: Istanbul University, Faculty of Health Science, Division of Physiotherapy and Rehabilitation
Brief Title: The Effects of Kinesio Tape Application With Different Verbal Input Given to With Patients With Rotator Cuff Tear
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University (Other)
Responsible Party: Principal Investigator, Yıldız Analay Akbaba, Assist Prof., Istanbul University
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Other
Other Study IDs: IU
Record Dates: First submitted 2017-01-12; First posted 2017-03-08 (Actual); Last update posted 2017-03-13 (Actual); Status verified 2017-03

CONDITIONS: Rotator Cuff Tear
Keywords: shoulder pain; shoulder function
MeSH Terms: conditions — Rotator Cuff Injuries; Shoulder Pain

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Group 1 (Experimental): it has been limited evidence of KT is effective
  Interventions: Other: Negative Verbal Input
- Group 2 (Experimental): it has been not known that KT is effective or not
  Interventions: Other: Neutral Verbal Input
- Group 3 (Experimental): it has been known that KT has excellent result
  Interventions: Other: Positive Verbal Input

INTERVENTIONS:
Other: Negative Verbal Input — The treatment group received a standardized therapeutic KT application. The physical therapist said that it has been limited evidence of KT is effective during application.
  Arms: Group 1
Other: Neutral Verbal Input — The treatment group received a standardized therapeutic KT application. The physical therapist said that it has been not known that KT is effective or not during application.
  Arms: Group 2
Other: Positive Verbal Input — The treatment group received a standardized therapeutic KT application. The physical therapist said that it has been known that KT has excellent result during application.
  Arms: Group 3

SUMMARY:
The aim of the study to investigate the effectiveness KT application with different verbal inputs on pain, function and range of motion (ROM) on patient with rotator cuff tear.

DETAILED DESCRIPTION:
Rotator cuff tears are most common of shoulder pain and functional limitations. Kinesio tape (KT) are frequently used in the conservative treatment of shoulder pathology. Even if some studies showed that KT is effective on pain, we think that it is due to positive thoughts of the patients about KT. The aim of the study to investigate the effectiveness KT application with different verbal inputs on pain, function and range of motion (ROM) on patient with rotator cuff tear. 97 patients (Group 1, n=32; Group 2, n=33, Group 3, n=32) were randomized into 3 groups according to verbal input given to patients about the effectiveness of KT; Group 1 (it has been limited evidence of KT is effective), Group 2 (it has been not known that KT is effective or not), Group 3 (it has been known that KT has excellent result). The same standard KT was applied to 3 groups. The rest, night and pain in activity were assessed by Visual Analog Pain Scale (VAS) before, after 30 min and 24 hours after KT application. ROM assessed by goniometer and the function was evaluated by Disabilities of the Arm, Shoulder and Hand (DASH) and the American Shoulder and Elbow Surgery score (ASES) before and 24 hours of KT application. Minimal clinically important difference and effective were calculated for the assessments used in the study.

ELIGIBILITY:
Inclusion Criteria:

* Patients were included in the study if they had a partial rotator cuff tear diagnosed on clinical grounds
* No episodes of shoulder instability
* No radiographic signs of fracture of the glenoid or the greater or lesser tuberosity MRI evidence of cuff tear
* Duration of symptoms of at least 3 months,
* Inadequate response to nonoperative management (including nonsteroidal anti-inflammatory drugs, physical therapy, rest, and 1 local corticosteroid injection) Positive empty can test indicating possible supraspinatus involvement
* Positive Hawkins-Kennedy test indicating possible external impingement, -Subjective complaint of difficulty performing activities of daily living
* 20 to 50 years of age.

Exclusion Criteria:

* Patients were excluded from the study if they had inflammatory joint disease -Rheumatologic disease Osteoarthritis of humerus head
* Prior surgery on the affected shoulder
* Inability to complete questionnaires because of language problem or cognitive disorder
* Shoulder girdle fracture
* Glenohumeral dislocation/subluxation
* Acromioclavicular sprain
* Concomitant cervical spine symptoms
* A history of shoulder surgery
* Patients who did not accept to participate
* Patients who did not come to the second evaluation.

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 87 (Actual)
Dates: Start 2016-01; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Visual Analogue Scale | The rest, night and pain in activity were assessed by VAS before and after 30 min, before and after 24 hours of KT application
  Pain intensity was assessed using the VAS; each patient was asked the pain during the rest, activity, and at night (on a 0 -10 numerical pain rating scale with zero corresponding to no pain and 10 corresponding to terrible pain). The rest, night and pain in activity were assessed by VAS before, after 30 min and 24 hours after KT application

SECONDARY OUTCOMES:
Shoulder range of motion | ROM (range of motion) assessed by goniometer before and 24 hours of KT application.
  Shoulder ROM measurements of forward flexion, abduction, and scapular plane external -internal rotation were taken using a standard goniometer. Pain-free active ROM and passive ROM were assesment.
Disabilities of the Arm, Shoulder and Hand questionnaire | Disabilities of the Arm, Shoulder and Hand (DASH) was evaluated before and 24 hours of KT application.
  The Disabilities of the Arm, Shoulder and Hand questionnaire is a 30-item scale of disability symptoms used to assess a patient's health status. The scores obtained from all items are then used to calculate a score ranging from 0 (no disability) to 100 (most severe disability).Disabilities of the Arm, Shoulder and Hand (DASH) was evaluated before and 24 hours of KT application.
American Shoulder and Elbow Surgery score (ASES) | American Shoulder and Elbow Surgery score was evaluated before and 24 hours of KT application.
  The ASES (American Shoulder and Elbow Surgery score) consists of 2 sections: a patient self-evaluation component and an assessment performed by a physician. The patient self-evaluation section has 11 items that can be used to generate a score. These items are divided into 2 areas: pain (1 item) and function (0 items). The function questions ask patients whether they can perform 10 daily life activities. Additionally, they are asked whether they can do their usual work and take part in normal sporting activity. Scores on the ASES range from 0 (absence of function) to 100 (normal function). The four-point Likert scale for the function questions ranges from 0 (unable to do) to 3 (not hard). American Shoulder and Elbow Surgery score was evaluated before and 24 hours of KT application.

IPD SHARING:
Plan to Share IPD: Yes